CLINICAL TRIAL: NCT01019018
Title: Efficacy of Subtenon Anesthesia With Olive Tipped Cannula: a Randomized Controlled Trial
Brief Title: Efficacy of Subtenon's Block With Olive Tipped Cannula
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Khaled Eye Specialist Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RP 0928
Record Dates: First submitted 2009-11-17; First posted 2009-11-25 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2009-11

CONDITIONS: Cataract
Keywords: subtenon block
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stevens cannula (Active Comparator): Subtenon with stevens cannula
  Interventions: Device: subtenon block
- Olive tip (Experimental): Olive tip group
  Interventions: Device: subtenon block

INTERVENTIONS:
Device: subtenon block — subtenon block with stevens cannula
  Arms: Stevens cannula
Device: subtenon block — subtenon block with Olive tip cannula cannula
  Arms: Olive tip

SUMMARY:
The purpose of this study is to compare the efficacy of olive tip cannula to the standard Steven's cannula in performing subtenon's anesthesia for patients undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing cataract extraction procedure under local anesthesia

Exclusion Criteria:

* Patients allergic to local anesthetic solutions.
* Presence local sepsis,
* Previous retinal or strabismus surgery in the same eye.
* Orbital abnormalities
* Previous subtenon's block in the same quadrant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Measurement of Akinesia score | 10 minutes after the block

SECONDARY OUTCOMES:
Surgeon satisfactions score | At the end of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- king Khaled Eye Specialist hospital, Riyadh, Saudi Arabia